CLINICAL TRIAL: NCT03262545
Title: Efficacy and Safety of Apatinib As Third Line Therapy in Patients With Advanced Ovarian Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sichuan Cancer Hospital and Research Institute (Other)
Responsible Party: Principal Investigator, Mei Kai, associate senior doctor, Sichuan Cancer Hospital and Research Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Ahead-OV-201704
Record Dates: First submitted 2017-08-22; First posted 2017-08-25 (Actual); Last update posted 2017-08-28 (Actual); Status verified 2017-08

CONDITIONS: Angiogenesis Inhibitors，Ovarian Neoplasms
MeSH Terms: interventions — apatinib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): apatinib 500 mg p.o. once daily
  Interventions: Drug: apatinib
- control group (Placebo Comparator): placebo p.o. once daily
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: apatinib — Patients in experimental group will take 500mg apatinib daily orally，and patients in control group will take placebo
  Arms: experimental group
Drug: Placebos — Physical properties of placebos are consistent with apatinib
  Arms: control group

SUMMARY:
The study is to investigate the efficacy and safety of apatinib in patients with advanced ovarian cancer,who has received second-line chemotherapy and failed.

DETAILED DESCRIPTION:
Ovarian cancer is the third most common gynecological malignancy，just less than endometrial cancer and cervical cancer. Because most patients with advanced ovarian cancer can not get the ideal tumor cell reduction surgery, and multi-drug resistance often emerges after repeated chemotherapy，recurrent and metastatic ovarian cancer has become one of the major diseases that threaten women's health. There is strongly necessary to explore effective therapeutic drugs and means to improve prognosis of these patients and improve the quality of life. The study，as a double blind clinical trial ,is to investigate the efficacy and safety of apatinib in patients with advanced ovarian cancer,who has received second-line chemotherapy regimens and failed. A total of 60 patients with performance status 0-2 were enrolled in this study, and were randomly divided into two groups--one group of 40 patients receiving apatinib，and another of 20 patients receiving placebo.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years to 70 years;
2. Had a histologically or cytologically confirmed diagnosis of epithelial ovarian cancer；
3. unfit for radical surgery and had received second-line chemotherapy，the disease still progressed or can not tolerate the chemotherapy;
4. Had a disease status that was measurable or evaluable as defined by Response Evaluation Criteria in Solid Tumors (RECIST, version1.1);
5. Had an Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0, 1, or 2;
6. Had a life expectancy of at least 12 weeks;
7. Adequate hepatic, renal, heart, and hematologic functions (hemoglobin ≥90g/L, platelets ≥ 80×10^9/L, neutrophils ≥ 1.5×10^9/L, total bilirubin within 1.5×the upper limit of normal (ULN), and b) ALT and AST≤2.5×the ULN (If liver metastases, serum creatine ≤ 1.5 x ULN);
8. Had not gastrointestinal diseases that lead to malabsorption or impact Drug absorption;
9. had good compliance;
10. Signed and dated informed consent.

Exclusion Criteria:

1. patients who had received anti-vascular therapy;
2. Allergic to any ingredients of Apatinib;
3. Participated in other drug clinical researchers within four weeks;
4. Have a variety of factors that affect oral medication (such as can not swallow, gastrointestinal resection, chronic diarrhea and intestinal obstruction, etc.)
5. Severe infection;
6. Patients with serious cardiovascular diseases,such as unstable angina, grade 3-4 heart dysfunction (NYHA Standard), congestive heart failure, poor-controlled arterial hypertension despite standard medical management;
7. Patients who received major surgical operations within 4 weeks before screening;
8. Patients who manifested arterial/venous thrombus events, e.g.cerebrovascular accident (including transient ischemic attack), deep venous thrombosis and pulmonary embolism, etc., within 12 months before screening;
9. Past or concurrent with other malignancies, except for cured skin basal cell carcinoma and cervical in situ cancer;
10. Have a history of psychiatric abuse and can not quit or have mental disorders.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-08-27 (Estimated); Primary Completion 2020-08 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | approximately 2 years
  Time from randomization until disease progression or death

SECONDARY OUTCOMES:
Overall survival (OS) | approximately 2 years
  Time from randomization until death from any cause of death
Objective response rate (ORR) | approximately 2 years
  Proportion of patients with reduction in tumor burden of a predefined amount
disease control rate (DCR) | approximately 2 years
  the total proportion of patients who demonstrate a response to treatment
Quality of life (QoL) | approximately 2 years
  As measured by the European Organization for Research and Treatment of Cancer questionnaire (EORTC QLQ C30)

CONTACTS AND LOCATIONS:
Locations (1):
- Sichuan Cancer Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gaitskell K, Rogozinska E, Platt S, Chen Y, Abd El Aziz M, Tattersall A, Morrison J. Angiogenesis inhibitors for the treatment of epithelial ovarian cancer. Cochrane Database Syst Rev. 2023 Apr 18;4(4):CD007930. doi: 10.1002/14651858.CD007930.pub3. PMID 37185961